CLINICAL TRIAL: NCT03036020
Title: The Norwegian Acute Stroke Prehospital Project
Acronym: NASPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristi G. Bache, PhD (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kristi G. Bache, PhD, Head of Research Department at The Norwegian Air Ambulance Foundation, Norwegian Air Ambulance Foundation
Organization: Norwegian Air Ambulance Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NASPP-2
Record Dates: First submitted 2014-12-01; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Acute Stroke; Traumatic Brain Injury
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contraindication anesthesiologists (Experimental): Ability of anesthesiologists to detect contraindications to thrombolysis in acute stroke patients prehospital by interpretation of prehospital cerebral CT scans
  Interventions: Radiation: CereTom Neurologica Samsung

INTERVENTIONS:
Radiation: CereTom Neurologica Samsung — Diagnosis of acute stroke patients by cerebral CT diagnostics prehospital

SUMMARY:
The main aim of the NASPP study is to assess the efficacy and safety of the prehospital diagnosis of stroke using the Norwegian stroke ambulance concept. NASPP aims to demonstrate that anesthesiologists trained in pre-hospital critical care may perform acute stroke diagnostics by clinical assessment and CT scan interpretation and integrating these skills in the already existing organizational frame of the Norwegian prehospital EMS system.

NASPP will systematically explore the Norwegian model of prehospital acute stroke diagnostics prior to the implementation of prehospital thrombolytic stroke treatment. NASSP will equip a regular ambulance staffed with a specially trained anesthesiologist and a specialized nurse. NASPP will perform the clinical part of the study in close co-operation with Østfold Hospital, Fredrikstad.

DETAILED DESCRIPTION:
Background Stroke is the third leading cause of death in most western countries, and the major cause of adult disability leaving two thirds of stroke survivors struggling with moderate to severe disability. Stroke affects approximately 15 million people worldwide each year.

Up to 90% of all strokes are ischemic (cerebral infarction), mostly due to an acute thromboembolic obstruction of a cerebral artery, whereas around 10 % of strokes are cerebral hemorrhages. Acute ischemic stroke must be considered as a medical emergency, and early recanalization of the obstructed artery must be attempted. The intravenous drug alteplase (Actilyse®), a recombinant human tissue type plasminogen activator, is approved for use within 4.5 hours after symptom start of an ischemic stroke. The earlier treatment is initiated, however, the better odds for of a good outcome.

A cerebral infarction cannot be differentiated from a cerebral hemorrhage without neuroradiological investigation. If a patient with acute cerebral hemorrhage is treated with thrombolysis it may be fatal. Therefore, and contrary to the setting of a cardiac infarction, intravenous thrombolysis of cerebral infarction has to be performed in-hospital after computer tomography (CT), or magnetic resonance imaging (MRI), scanning of the brain. The consequence of this obligatory radiological examination is an unavoidable time delay and very few ischemic stroke patients are actually treated within "the golden 90 minutes" after symptom onset. The only way to avoid this, for the brain, detrimental time delay is logical; to establish the diagnosis of ischemic stroke outside the hospital and in time as near symptom onset as possible. Subsequently this will open the possibility for very early prehospital thrombolytic treatment for a much higher number of patients.

Minimizing prehospital time delay has been proven to positively influence thrombolytic rates in acute ischemic stroke. However, a recent study with a telemedicine-equipped ambulance (telestroke ambulance) has shown that prehospital real-time stroke severity assessment by hospital-based stroke physicians during ambulance transport does not have a technical acceptable stability for clinical use. In this Berlin study using "actor stroke patients" in a moving ambulance, an acceptable clinical evaluation of only 40% of the patients was achieved. A recent clinical stroke study from the University Saarland, Germany has, however, demonstrated that the concept of prehospital stroke diagnosis is feasible. Using a specially designed mobile stroke unit (MSU), a car ambulance equipped with a stroke neurologist, a CT scanner and a point of care biochemical laboratory, time from symptom onset to diagnostic therapeutic decision for thrombolysis was reduced from 76 to 35 minutes. The CT scanner in the MSU was shown to provide brain scans of high quality in 95% of cases allowing differentiation of cerebral infarction and cerebral hemorrhage. No safety radiation issues occurred for either staff or patients.

The time delay in stroke diagnostics may be reduced with early radiological diagnosis, but there is also need of reliable clinical recognition of stroke symptoms. The reliability of the National Institutes of Health Stroke Scale (NIHSS) is established by several clinical trials when performed by trained neurologists. Dewey et al proved in a 1999 trial "Inter-rater reliability of the National Institutes of Health Stroke scale: Rating by Neurologists and Nurses in a Community-Based stroke Incidence study" that the overall agreement in NIHSS scoring between trained nurses and a trained neurologists were no different from the agreement between neurologists. The study suggested that trained nurses could administer the NIHSS with reliability similar to stroke- trained neurologists.

Aims The main aim of the NASPP study is to assess the efficacy and safety of the prehospital diagnosis of stroke using the Norwegian stroke ambulance concept. NASPP aims to demonstrate that anesthesiologists trained in pre-hospital critical care may perform acute stroke diagnostics by clinical assessment and CT scan interpretation and integrating these skills in the already existing organizational frame of the Norwegian prehospital EMS system.

NASPP will systematically explore the Norwegian model of prehospital acute stroke diagnostics prior to the implementation of prehospital thrombolytic stroke treatment. NASSP will equip a regular ambulance staffed with a specially trained anesthesiologist and a specialized nurse. NASPP will perform the clinical part of the study in close co-operation with Østfold Hospital, Fredrikstad.

Hypothesis Cerebral CT examination by an anesthesiologist trained in prehospital care; feasible and accurate after a stroke? An anesthesiologist trained in pre-hospital care will be able to perform, assess and transfer by teleradiology cerebral CT scans from patients presenting with stroke symptoms lasting no more than 4 hours. The performance of the anesthesiologists will be compared to independent assessments may by a radiologist or a neurologist at the admission hospital, and further on with a neuroradiologist.

The prehospital diagnosis of ischemic stroke by an anesthesiologist trained in prehospital critical care - a new concept. An anesthesiologist trained in pre-hospital critical care will make an accurate prehospital clinical and radiological diagnosis of acute ischemic stroke, enabling early prehospital thrombolytic treatment.

Long-term prognostic value of NIHSS assessment in the prehospital phase of ischemic stroke. To assess if a prehospital NIHSS score may predict long-term (3 months) patient outcome assessed with the modified Rankin Scale (mRS), in acute stroke patients treated or not treated with thrombolysis.

Design NASPP is an observational and cross-sectional study, designed to test the efficiency and accurancy of prehospital diagnostics of acute stroke in a Norwegian stroke ambulance concept. NASPP is considered a pilot study, due to paucity of data in the literature and lack of existing medical experience. NASPP will aim to include up to 200 patients.

Methods and material: Clinical study Cerebral CT examination by an anesthesiologist trained in prehospital care; feasible and accurate after a stroke? Prehospital ischemic stroke diagnostics by an anesthesiologist trained in prehospital critical care - a new concept.

After completing a preclinical study we aim to prove that anesthesiologists trained in pre-hospital critical care can perform "state of the art" prehospital acute stroke diagnostics. Patient care delivery will be conducted in a specially designed stroke ambulance operating from Østfold Hospital, Fredrikstad. The stroke ambulance will respond to all patients over the age of 18 in contact with 113 emergency dispatch center presenting symptoms of paresis of arm and or legs, facial paresis, visual or speech disturbances (Norwegian Index of medical emergencies chapter 27.03-27.05). The local dispatch center will send the stroke ambulance for an emergency turnout to the patient. The stroke ambulance will operate from 08.00 am to 20.00 p.m. during weekdays in the study period, because of practical and economical considerations. The stroke ambulance will only respond to patients localized more than 10 -15 minutes drive from the hospital, to make sure that no time is lost to those living in the very close proximity to the hospital. The dispatch center will simultaneously alarm the on-call neurologist at Østfold Hospital, Fredrikstad.

The Norwegian Air Ambulance Foundation will organize the training of the stroke ambulance crew (anesthesiologist and nurse trained in prehospital care). The training course is based on the preclinical trail, and also including simulation training in the stroke ambulance. The ambulance anesthesiologist will complete a test in interpretation of cerebral CT scans in acute stroke, and a NIHSS certification. The anesthesiologist and the nurse will both be trained to operate the biochemical point of care laboratory (glucose, platelets, INR and Hb) and the CT machine.

The stroke ambulance will respond to all patients with stroke symptoms meeting the inclusion criteria. A total of 400 patients will be included, and all patients will be asked for oral consent. If aphasic, or having reduced consciousness, the patient will be included in the study. On site the anesthesiologist will do a rapid screening using the ABCDE's of trauma care. If the patient is stable and further investigations can proceed the NIHSS score will be completed. The patient will get two venous lines, and blood samples will be collected. Blood samples for GFAP and S-100 B will be stored and delivered to the laboratory at the hospital for further analyses. A circulatory stabile patient will be taken into the stroke ambulance, were the CT scan can be performed. In circulatory unstable patients the ambulance anesthesiologist can decide not to perform the CT scan but head directly to the hospital.

While the CT scan is taken the blood samples are analyzed in the point of care laboratory. The ambulance anesthesiologist assesses the CT scan and fills out the study forms. The CT scan is simultaneously sent to Østfold Hospital, Fredrikstad for interpretation by the neurologist and the radiologist on call. The patient transport to the hospital and the communication with the neurologist on call will follow standard procedures. The anesthesiologist will not report the results of NIHSS score or CT scans, as the study form completed by the anesthesiologist is for research purpose only. The ambulance anesthesiologist will be medically responsible for the patient until hospitalization. The neurological team on call will provide further medical care, and if appropriate start thrombolytic treatment after patient admission.

A neuroradiologist will, without any clinical knowledge, review the CT scans after the study has included at least 400 patients. The results from the initial interpretation by the ambulance anesthesiologist are held anonymous, and blinded for the neuroradiologist. The in-hospital written reports will be collected and reviewed. The results will be analyzed statistically to show distribution of the different categories of inter-rater agreement, compared to the neurologists and radiologists at the admission hospital.

To test hypothesis the anesthesiologist trained in pre-hospital critical care will decide upon whether he/she would have given thrombolytic treatment to the patient based upon clinical findings, anamnestic information, NIHSS score, laboratory test results and CT scan interpretation. Therapy decision will only be written in the study form, and not reported to the hospital. Retrospectively the therapy decision made by the anesthesiologist will be statistically compared to the therapy decision made by the in-hospital stroke team. We aim to determine the level of inter-rater agreement between the stroke anesthesiologist and the in-hospital stroke team, with regard to their decision on thrombolysis and diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* All patients met by emergency services within 4 hours after symptom onset
* Stroke symptoms: sudden weakness of leg or arm, especially on one side, facial asymmetry and/or sudden trouble walking, and speech disturbance (Norwegian Index of medical emergencies 27.03-27.05).
* Patients from the Hospital dispatch center area, being more than 10-15 minutes drive from the hospital.
* Giving informed consent, written or oral, if possible or consent from relative at site

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Female < 50 years and uncertainty of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Inter-rated agreement between the anesthesiologist and the inhospital stroke team (radiologist and neurologist) | Baseline
  The ambulance anesthesiologist assesses the pre-hospital cerebral CT scan and fills out the predefined variables in designated study forms. All cerebral CT interpreations are categorized in 1) no radiological contraindication to thrombolytics 2) yes radiological contraindication to thrombolytics. The CT scan is simultaneously sent to the hospital, for interpretation by the neurologist and the radiologist on call. The anesthesiologist intgerpration is blinded to the stroke team. A neuroradiologist will, without any clinical knowledge, review the CT scans after the study has included is completed. The results from the initial interpretation by the ambulance anesthesiologist are held anonymous, and blinded for the neuroradiologist. The results will be analyzed statistically to show distribution of the different categories of inter-rater agreement, compared to the neurologists and radiologists at the admission hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Christian G Lund, MD Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Østfold Hospital Norway, Fredrikstad, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hov MR, Ryen A, Finsnes K, Storflor J, Lindner T, Gleditsch J, Lund CG; on behalf of the NASPP Group. Pre-hospital ct diagnosis of subarachnoid hemorrhage. Scand J Trauma Resusc Emerg Med. 2017 Feb 28;25(1):21. doi: 10.1186/s13049-017-0365-1. PMID 28245880